CLINICAL TRIAL: NCT01533467
Title: Study of Perineal Protection Device
Brief Title: A Device Designed to Protect the Perineum During Labor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Helsingborgs Hospital (Other)
Collaborators: Lund University Hospital (Other); Skane University Hospital (Other)
Responsible Party: Principal Investigator, Knut Haadem, Principal investigator, Helsingborgs Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KH-HBG-12; 148/2008 (Other Grant/Funding Number: Thelma Zoegas and Stig och Ragna Gortons Foundation)
Record Dates: First submitted 2012-02-06; First posted 2012-02-15 (Estimated); Last update posted 2012-02-15 (Estimated); Status verified 2012-02

CONDITIONS: Perineal Tear
Keywords: Delivery rupture; perineal protection device; reduce perineal tears

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Perineal device used (Other): Use of the perineal device during delivery
  Interventions: Device: Perineal protection device
- No intervention (No Intervention): Controls, delivered as normal

INTERVENTIONS:
Device: Perineal protection device — Use of the device during delivery and inspection afterwards to see the tears.
  Other Names: Manufacturer; Calle Gejde AB, 234 21 Lomma, Sweden
  Arms: Perineal device used

SUMMARY:
Objective:

To investigate the protective effects of a newly invented device for reducing tears in the perineum during vaginal childbirth.

Design:

A multicenter randomized control trial performed at three hospitals in Sweden, in Helsingborg, Lund and Malmö. Participants recruited are women with vaginal delivery (N=1200), cephalic presentation. They will be randomized to an intervention group, with a perineal protection device, and a control group deliver as normal.

Main outcome measures:

The effect on the frequency and extension of perineal ruptures grade I, II and anal sphincter rupture are measured.

DETAILED DESCRIPTION:
Perineal rupture shall be measured with a ruler. Anal sphincter ruptures be examined by physicians. Drawing be made of the tears by the midwife.

ELIGIBILITY:
Inclusion Criteria:

* Vaginal delivery

Exclusion Criteria:

* Age below 18 years and no understanding of written and oral information.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1200 (Actual)
Dates: Start 2010-11; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Grade I and II rupture during delivery | time at the delivery department (up to 12 months)
  Number and extension of perineal tears during delivery

CONTACTS AND LOCATIONS:
Overall Officials: Knut Haadem, MD, PhD, Principal Investigator — Dept Obstet & Gynecol, Helsingborg Hospital, Helsingborg, Sweden
Locations (1):
- Knut Haadem, Helsingborg, Helsingborg, Sweden

REFERENCES:
- [Derived] Lavesson T, Griph ID, Skarvad A, Karlsson AS, Nilsson HB, Steinvall M, Haadem K. A perineal protection device designed to protect the perineum during labor: a multicenter randomized controlled trial. Eur J Obstet Gynecol Reprod Biol. 2014 Oct;181:10-4. doi: 10.1016/j.ejogrb.2014.07.006. Epub 2014 Jul 30. PMID 25126978